CLINICAL TRIAL: NCT02668289
Title: Periodontal Phenotype and Supracrestal Soft Tissue Dimentions - Clinical Correlations and Their Impact on Post-extraction Volumetric Changes
Brief Title: Periodontal Phenotype Study (Tooth Extraction)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gustavo Avila-Ortiz DDS, MS, PhD (Other)
Responsible Party: Sponsor-Investigator, Gustavo Avila-Ortiz DDS, MS, PhD, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201510790
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Tooth Extraction Status Nos
MeSH Terms: interventions — Consent Forms; Mass Screening; X-Rays; Moire Topography; Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- interventional (Other): consent, screening, xrays, PVS impressions, photographs, CBCT, anesthesia, extraction, clinical measurements
  Interventions: Other: consent; Other: Screening; Other: Xray; Other: PVS Impressions; Other: Photographs; Other: CBCT; Other: Anesthesia; Procedure: Extraction; Other: Clinical measurements

INTERVENTIONS:
Other: consent — At the initial screening examination, each subject will receive an informed consent form. Prior to signing the informed consent, one of the investigators or qualified staff will thoroughly discuss participation in the study with each subject, allocating time for questions and answers.
Other: Screening — At the initial screening examination, complete medical and dental history will be obtained to verify eligibility.
Other: Xray — each subject will undergo site-specific oral radiographic exam (new periapical radiographs will be obtained if needed) to evaluate potential study sites.
Other: PVS Impressions — PVS impressions of the arch of interest will be obtained in order perform volumetric analysis of the area of interest.
Other: Photographs — Intraoral photographs will also be taken and subsequent study visits will be planned.
Other: CBCT — The patient will then be sent to the Department of Radiology at the College of Dentistry for a baseline CBCT and follow-up at 14 week CBCT. These CBCT's will be utilized to evaluate the hard tissue volume in comparison to the clinical volume of soft tissue.
Other: Anesthesia — After appropriate local anesthetic is administered and anesthesia is achieved, the buccal tissue thickness will be measured and recorded.
Procedure: Extraction — After the pre-extraction baseline measurements are recorded and adequate anesthesia is confirmed, minimally invasive extraction procedures will be initiated. All extractions will be performed by residents in the UI CoD Periodontics advanced education program.
Other: Clinical measurements — Measuring soft tissue dimensions, bone thickness prior to and immediately after extraction and then after appropriate healing time frames.

SUMMARY:
The purpose of this trial is to determine the correlations between various tissue dimensions and the changes that occur following a single-tooth dental extraction in human adults.

65 adult subjects who are in need of dental extractions will be recruited. Clinical measurements will be gathered prior to and immediately following the single tooth extraction. There will be a 2-week post-operative visit to assess healing and a 14-week follow-up for photographic documentation and clinical measurements of the extraction area.

DETAILED DESCRIPTION:
Periodontal phenotype, also known as periodontal biotype, has been recognized as one of the key factors that may potentially impact the outcome of a variety of esthetic restorative procedures. With the increasing esthetic demand of patients in the context of tooth replacement therapy in the anterior esthetic zone, the ability to determine the prognostic value and the influence on treatment outcomes of this parameter has become a critical component of contemporary treatment planning. Periodontal phenotype encompases "bone morphotypes, shapes of the teeth, morphologic characteristics of the gingiva and the periodontium".

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75 years
* Gender: No restriction
* Subjects must require a single-rooted tooth extraction (Tooth deemed as periodontally and/or restoratively hopeless) in the maxillary anterior region (first premolar to first premolar)
* Subjects must be able and willing to follow instructions related to the study procedures
* Subjects must have read, understood and signed an informed consent form

Exclusion Criteria:

* More than 1 mm of recession present on the tooth planned for extraction and inclusion in the study
* Reported allergy or hypersensitivity to any of the products to be used in the study
* Severe hematologic disorders, such as hemophilia or leukemia
* Active severe infectious diseases that may compromise normal healing
* Liver or kidney dysfunction/failure
* Currently under cancer treatment or within 18 months from completion of radio- or chemotherapy
* Subjects who have a long-term history of oral bisphosphonate use (i.e. 10 years or more)
* Subjects with a history of IV bisphosphonates
* Subjects with uncontrolled diabetes, defined as Hba1c > 7.0
* Subjects with severe metabolic bone diseases, such as Paget's disease of bone, will be excluded
* Pregnant women or nursing mothers
* Heavy smokers: Subjects who have smoked >10 cigarettes per day within 6 months of study onset
* Concomitant medications: Subjects on concomitant drug therapy for systemic conditions that may affect the outcomes of the study will not be included in the study.

NOTE: Occasional, short-term use (7-14 days) of analgesics or common cold medications is permitted. Use of such medications will be reviewed and recorded by the investigator.

- Any other non-specified reason that from the point of views of the investigators will make a candidate not a suitable subject for the study (e.g. limited mouth opening).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-01-31 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Percentage change in tissue volume - Rank Correlations | 14 weeks
  For the purpose of this study, a 10-20% reduction in the volume must detectable. Pearson correlations will be used to assess associations if appropriate and Spearman rank correlations will be considered if needed.

SECONDARY OUTCOMES:
Probing Depths of soft tissue dimensions | 14 weeks
  supracrestal soft tissue dimensions will be evaluated
bone thickness ( facial and lingual) - Correlations | 14 weeks
  Analogous correlational approaches, supplemented by regression methods, will be used to assess the relationships between measurements made by CBCT with those derived from volumetric analysis of casts.
soft tissue thickness (facial and lingual) -correlations | 14 weeks
  correlations among the periodontal phenotype and the supracrestal soft tissue dimensions will be evaluated.

OTHER OUTCOMES:
width of keratinized gingiva | 14 weeks
  supracrestal soft tissue dimensions will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Avila Ortiz, BSE, DDS, Principal Investigator — University of Iowa
Locations (1):
- UIowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Couso-Queiruga E, Graham ZA, Peter T, Gonzalez-Martin O, Galindo-Moreno P, Avila-Ortiz G. Effect of periodontal phenotype characteristics on post-extraction dimensional changes of the alveolar ridge: A prospective case series. J Clin Periodontol. 2023 May;50(5):694-706. doi: 10.1111/jcpe.13781. Epub 2023 Feb 1. PMID 36644815